CLINICAL TRIAL: NCT03956199
Title: Managing Irreversible Pulpitis - The Effectiveness of Pulpotomy Compared to Root Canal Treatment as a Replacement for Conventional Root Canal Treatment: A Multicentre Randomized Controlled Trial
Brief Title: Pulpotomy vs.Root Canal Treatment in Managing Irreversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PB-PG-0817-20040
Record Dates: First submitted 2019-05-14; First posted 2019-05-20 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Pulpitis - Irreversible
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental pulpotomy (Experimental)
  Interventions: Procedure: pulpotomy
- Root canal treatment (Active Comparator)
  Interventions: Procedure: Root canal treatment

INTERVENTIONS:
Procedure: pulpotomy — removal of the pulp from pulp chamber
  Arms: experimental pulpotomy
Procedure: Root canal treatment — Removal of at the entire content of the root canal system and root canal obturation
  Arms: Root canal treatment

SUMMARY:
The study aims to compare two methods of repairing and saving a badly damaged or infected tooth. One method is called root canal treatment (RoCT) and the other (new method) is called pulpotomy. RoCT involves removing the damaged area of the tooth including the tooth nerve (called the pulp), cleaning, disinfecting and sealing it. Pulpotomy however attempts to preserve as much of the tooth nerve as possible (keeping the tooth alive). RoCT is more expensive and painful. Therefore, some patients delay or avoid getting treated, resulting in later complications treated in an emergency setting. This research will aim to show that pulpotomy is less painful, less involved (i.e. less invasive), less time consuming and consequently more cost effective. Long term costs of dental treatment as well as the improved quality of life will therefore offer benefits for patients, public and the NHS who use dental services. Caries (tooth decay) is the most common diseases in the world. The NHS spends at least £3.4 billion per year on dental visits or at dental hospitals. This does not include private (societal) costs to individuals who do not qualify for NHS dental treatment. Consequently, those who end up avoiding or delaying treatment result in complications often treated through the NHS. We have therefore chosen a randomized controlled trial design, a gold standard method to compare the effectiveness of the two treatment options. The participants will be 168 dental patients (male or female) from different parts (London and Liverpool) of the UK so that results can be generalized. This design was considered in consultation with a member of the public (a co-applicant) who will be involved in the trial from the start to completion. The results will be published and discussed at conferences as well as through our patient and public network.

ELIGIBILITY:
Inclusion Criteria:

* • Dental patients from an acute (secondary care) setting from at least three UK centres (including King's College London Dental Institute, Denmark Hill and Liverpool).

  * Male or female (aged >16) able to provide informed consent in otherwise good general health with at least one molar tooth with clinical symptoms of irreversible pulpitis caused by caries, requiring RoCT (endodontic treatment).
  * Patients enrolled will have clinical symptoms of irreversible pulpitis who need treatment.

Exclusion Criteria: Exclusion Criteria:

* The presence of fistulas or swelling
* Anterior teeth or premolars
* External or internal root resorption
* Multiple teeth with carious lesions in the same quadrant,
* Pregnant women, in view of requirements for radiographs.
* Patients younger than 16.
* Patients unable to give consent.
* Patients who have been administered antibiotics in the previous month.
* Immunocompromised patients
* Teeth with hopeless prognosis with caries extended into root dentine and with tooth margin at crestal bone level

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Short term pain following pulpotomy versus root canal treatment | 7 days
  Pain, tenderness or swelling assessment at baseline and over the first 7 days post completion of treatment using a daily diary of pain (based on a 10 point visual analogue (VAS Scale), measured using the area under the curve (AUC) approach).

SECONDARY OUTCOMES:
Cost-effectiveness of pulpotomy | 2 years
  • Health care resource use between randomization and 12 months post randomization for assessing the cost-effectiveness of pulpotomy in comparison to RCT as measured by the incremental cost-effectiveness ratio (ICER) in terms of the INMB
sensitivity and specificity of CBCT versus periodical radiographs to detect periapical radiolucencies | 2 years
  the sensitivity and specificity of periapical radiograph (clinical standard) to CBCT (experimental) in terms of detection of periapical disease.
success rates of pulpotomy compared to root canal treatment | 2 years
  The vitality or absence of apical pathology of the tooth at 24 months: that is, an absence of either pain, swelling or tenderness to biting of the tooth and no evi-dence of inflammation in the tissues around the tip of the root detected by con-ventional radiographs and CBCT (independent assessors) after 24 months from randomisation. Both assessors must agree to conclude an overall absence of apical pathology. Treatment outcome will be assessed objectively using scans taken pre-treatment and and follow-up (6,12,24 months) appointments.
Quality of life difference between patients that receive pulpotomy versus root canal treatment | 12 months
  • The EQ-5D-3L and EQ-5D-5L measured at baseline, over the first 7 days, 6 and 12 months post randomisation. One major feature of the EQ-5D tool is that the health states obtained from the questionnaire may be con-verted into a single index value with country specific value sets. This will facilitate the calculation and comparison of quality-adjusted life years (QALYs) between pulpotomy vs. primary root canal treatment. The QALY is a measure of disease burden including the quality and quantity of life lived, with one QALY equating to one year in perfect health

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Royal Liverpool University Hospital, Liverpool
  - Guy's Hospital, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel N, Khan I, Jarad F, Zavattini A, Koller G, Pimentel T, Mahmood K, Mannocci F. The short-term postoperative pain and impact upon quality of life of pulpotomy and root canal treatment, in teeth with symptoms of irreversible pulpitis: A randomized controlled clinical trial. Int Endod J. 2025 Jan;58(1):55-70. doi: 10.1111/iej.14144. Epub 2024 Sep 26. PMID 39325552